CLINICAL TRIAL: NCT04838353
Title: Evaluation of the Safety and Effectiveness of a Percutaneously Created Interatrial Shunt to Alleviate Heart Failure Symptoms in Patients With Chronic Heart Failure and Preserved or Mid-Range Left Ventricular Ejection Fraction
Brief Title: Alleviate-HF-2 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alleviant Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0002
Record Dates: First submitted 2021-04-01; First posted 2021-04-09 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ALV1 System — The ALV1 system is designed to create a controlled size interatrial shunt via a proprietary intra-cardiac catheter. There is no temporary or permanent implant used to create or maintain the interatrial shunt. The therapy is intended to be delivered in a single procedure administered under general anesthesia in a cardiac catheterization laboratory.

SUMMARY:
Patients with heart failure and preserved left ventricular ejection fraction (HFpEF, EF ≥ 50%) or mid-range left ventricular ejection fraction (HFmrEF, 40% < EF < 50%) with mild to moderate functional limitation will be evaluated for treatment via creation of a no-implant interatrial shunt using clinical, echocardiographic, and invasive hemodynamic data

ELIGIBILITY:
Inclusion Criteria:

1. NYHA Class II at screening with a prior history of greater than NYHA Class II, OR NYHA Class III at screening, OR ambulatory Class IV at screening: with documented medical history of heart failure for at least 6 months prior to the screening visit.
2. Medical history within the past 12 months of at least one hospitalization with heart failure as the primary or secondary diagnosis OR treatment with IV diuretics for heart failure..
3. LVEF (by Echo) > 40% as measured by the study-specific transthoracic echocardiography.
4. Echocardiographic evidence of diastolic dysfunction documented by one or more of the following as measured by the study-specific transthoracic echocardiography protocol:

   1. LA diameter > 4cm
   2. LA volume index >28 mL
   3. Lateral e' <10 cm/s
   4. Septal e' <8 cm/s
   5. Lateral E/e' >10
   6. Septal E/e' >15
5. As measured by the study-specific exercise hemodynamic right heart catheterization protocol performed during screening: Elevated left atrial pressure WITH a gradient compared to right atrial pressure (RAP) documented by: (1) end-expiratory PCWP at peak supine cycle ergometer exercise ≥ 25mmHg AND (2) PCWP greater than RAP by ≥ 5 mmHg, OR (1) ≥ 10 mmHg increase of end-expiratory PCWP at peak supine cycle ergometer exercise compared to resting PCWP AND (2) PCWP greater than RAP by ≥ 5 mmHg. Patients must also have PCWP greater than RAP by ≥ 5 mmHg at rest.

Exclusion Criteria:

1. Presence of advanced heart failure defined as one or more of the following:

   * ACC/AHA/ESC Stage D heart failure, non-ambulatory NYHA Class IV HF.
   * Cardiac index less than 2.0 L/min/m2.
   * Patient is on the cardiac transplant waiting list.
   * Inotropic infusion (continuous or intermittent) for EF less than 40% within the past 6 months.
2. Presence of moderate or worse valve disease, defined as one or more of the following:

   * Moderate or worse mitral valve regurgitation or moderate or worse mitral stenosis.
   * Moderate or worse tricuspid valve regurgitation.
   * Moderate or worse aortic valve disease defined as moderate or worse AS or AI.
3. . Presence of chronic pulmonary disease defined by one or more of the following:

   * Requirement for continuous home oxygen use.
   * Hospitalization within the past 12 months for treatment of pulmonary disease.
   * Significant chronic pulmonary disease defined as FEV1 less than 50%.
4. Documented as currently requiring dialysis or estimated GFR less than 25ml/min/1.73m2
5. 6-minute walk distance less than 50 m or greater than 450 m performed during screening.
6. Documented atrial fibrillation with ventricular rate greater than 100 BPM at screening.
7. Presence of moderate or worse right heart dysfunction OR RV dysfunction defined as TAPSE less than 14 mm or RVFAC less than or equal to 30%
8. Presence of pulmonary hypertension with PASP greater than or equal to 70 mmHg OR PVR greater than 4 Wood units.
9. Presence of anatomic anomaly that precludes creation of interatrial shunt (including patent foramen ovale, atrial septal defect, target septal thickness greater than 3 mm)
10. SBP greater than 170 mmHg at screening.
11. Documented left ventricular end diastolic diameter greater than 6 cm.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The composite incidence of one or more major adverse cardiac, cerebrovascular and thromboembolic events and change in supine exercise PCWP at peak exercise. | At 1 month and through 12 months
  Defined as cardiovascular death, embolic stroke, embolic myocardial infarction, pulmonary or arterial embolism, device-and/or procedure-related serious adverse cardiac events.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (2):
  - Flinders Medical Centre, Adelaide
  - Monash Medical Centre, Clayton
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Canada
- Southern District Health Board, Dunedin, New Zealand
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Laufer-Perl M, Flint N, Arbel Y, Alenezi F, Kittipibul V, Yaranov D, Shaburishvili T, Amin R, Fudim M. Atrial Mechanics in Heart Failure With Preserved Ejection Fraction: Effect of a No-Implant Interatrial Shunt. Circ Heart Fail. 2025 Oct;18(10):e012573. doi: 10.1161/CIRCHEARTFAILURE.124.012573. Epub 2025 Sep 3. PMID 40899260
- [Derived] Udelson JE, Barker CM, Wilkins G, Wilkins B, Gooley R, Lockwood S, Potter BJ, Meduri CU, Fail PS, Solet DJ, Feldt K, Kriegel JM, Shaburishvili T. No-Implant Interatrial Shunt for HFpEF: 6-Month Outcomes From Multicenter Pilot Feasibility Studies. JACC Heart Fail. 2023 Aug;11(8 Pt 2):1121-1130. doi: 10.1016/j.jchf.2023.01.024. Epub 2023 Apr 26. PMID 37115132